CLINICAL TRIAL: NCT02057172
Title: A Phase II, 12-week, Double-blind, Randomised, Parallel Group, Multi-centre, International Trial to Assess the Effect on Glycaemic Control of Five Doses of HM11260C Versus Placebo or Open-label Liraglutide in Subjects With Type 2 Diabetes
Brief Title: Glycaemic Control of Weekly LAPS-Exendin Versus Placebo in Subjects of Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HM-EXC-203
Record Dates: First submitted 2014-01-30; First posted 2014-02-06 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes
Keywords: glycaemic control; HM11260C; placebo; safety; tolerability; type 2 diabetes mellitus; efficacy; T2DM; glycated haemoglobin (HbA1c); glycosylated haemoglobin (HbA1c); Glucagon-Like Peptide-1 (GLP-1) agonists; blood sugar levels; fasting plasma glucose (FPG)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- HM11260C (0.3 mg) (Experimental): Weekly administration of 0.3 mg of HMC11260C by subcutaneous injection for 12 weeks
  Interventions: Drug: HM11260C
- HM11260C (1 mg) (Experimental): Weekly administration of 1 mg of HM11260C by subcutaneous injection for 12 weeks
  Interventions: Drug: HM11260C
- HM11260C (2 mg) (Experimental): Weekly administration of 2 mg of HM11260C by subcutaneous injection for 12 weeks
  Interventions: Drug: HM11260C
- HM11260C (3 mg) (Experimental): Weekly administration of 3 mg of HM11260C by subcutaneous injection for 12 weeks
  Interventions: Drug: HM11260C
- HM11260C (4 mg) (Experimental): Weekly administration of 4 mg of HM11260C by subcutaneous injection for 12 weeks
  Interventions: Drug: HM11260C
- Placebo (Placebo Comparator): Weekly administration of placebo by subcutaneous injection for 12 weeks
  Interventions: Drug: Placebo
- Liraglutide (Active Comparator): Liraglutide will be administered daily, at doses of 0.6 mg to 1.8 mg.
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: HM11260C — HM11260C is a novel long-acting form of CA Exendin-4 (an Exendin-4 analogue)
  Other Names: LAPS-Exendin-4
  Arms: HM11260C (0.3 mg); HM11260C (1 mg); HM11260C (2 mg); HM11260C (3 mg); HM11260C (4 mg)
Drug: liraglutide — Liraglutide is a GLP-1 agonist.
  Other Names: Victoza
  Arms: Liraglutide
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the optimal dose or doses of HM11260C, when administered once a week under the skin, to improve the control of blood sugar levels in patients with early-stage type 2 diabetes mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* Ages eligible for study : 18 years to 74 years
* Genders eligible for study : Male and Female
* Diagnosed with T2DM
* Received diet and exercise therapy with or without metformin monotherapy
* HbA1c levels of between ≥ 7.0% and ≤ 10.0%
* Females of childbearing potential who are not pregnant and agree to use a reliable method of birth control
* Written informed consent must be obtained

Exclusion Criteria:

* Pregnant or nursing (lactating) women
* Diagnosis of type 1 diabetes mellitus
* Uncontrolled diabetes defined as a FPG level of > 240 mg/dL
* A significant change in body weight in the 3 months before screening
* Any history of GI intolerance
* Personal or family history of medullary thyroid cancer (MTC) or a genetic condition that predisposes to MTC
* Known history of chronic pancreatitis
* A history of alcohol or drug abuse or drug addiction

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in baseline in glycosylated haemoglobin (HbA1c) at 12 weeks | Up to 127 days

SECONDARY OUTCOMES:
Fasting plasma glucose levels (FPG) | Up to 127 days
7-point glucose profile | Up to day 127
Other glycaemic control parameters | Up to day 127
Serum lipid profile | Up to day 127
Body weight | Up to day 127
Number of subjects attaining goal glycosylated haemoglobin (HbA1c) <7% | Up to 127 days

OTHER OUTCOMES:
Assess the safety and tolerability of HM11260C | Up to day 127
Assess the immunogenicity of HM11260C | Up to day 127

CONTACTS AND LOCATIONS:
Overall Officials: Hanmi Pharmaceutical, Study Director — clinical4@hanmi.co.kr
Locations (1):
- Hanmi pharmaceutical, CA, California, United States

REFERENCES:
- [Derived] Rosenstock J, Sorli CH, Trautmann ME, Morales C, Wendisch U, Dailey G, Hompesch M, Choi IY, Kang J, Stewart J, Yoon KH. Once-Weekly Efpeglenatide Dose-Range Effects on Glycemic Control and Body Weight in Patients With Type 2 Diabetes on Metformin or Drug Naive, Referenced to Liraglutide. Diabetes Care. 2019 Sep;42(9):1733-1741. doi: 10.2337/dc18-2648. Epub 2019 Jul 18. PMID 31320446